CLINICAL TRIAL: NCT07244393
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Preliminary Efficacy of Lutetium (177Lu) DGUL in Combination With Pembrolizumab in Patients With Metastatic Castration-Resistant Prostate Cancer (IGNITE Trial)
Brief Title: Lutetium (177Lu) DGUL Combined With Pembrolizumab in Metastatic Castration-Resistant Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cellbion Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lu-PSMAPem01; KEYNOTE-G28 (Other: Merck Sharp & Dohme LLC); MK-3475-G28 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — Lutetium; Lutetium-177; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Monotherapy Arm (Experimental): Monotherapy Arm: 10 patients will receive Lutetium (177Lu) DGUL monotherapy.
  Interventions: Drug: Lutetium (177Lu) DGUL
- Combination Arm (Experimental): Combination Arm: 20 patients will receive Lutetium (177Lu) DGUL in combination with pembrolizumab.
  Interventions: Drug: Lutetium (177Lu) DGUL; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lutetium (177Lu) DGUL — Lutetium (177Lu) DGUL will be administered in 4 doses at 6-week intervals (Q6W), and for patients showing good tolerance, additional 2 doses may be added, for a maximum of 6 doses.
Drug: Pembrolizumab — Pembrolizumab will be introduced at a dose of 400 mg every 6 weeks, beginning with the second cycle of Lutetium (177Lu) DGUL, and will continue for up to approximately 2 years (18 doses).
  Other Names: KEYTRUDA®
  Arms: Combination Arm

SUMMARY:
The goal of this clinical trial is to evaluate the safety of the combination therapy of Lutetium (177Lu) DGUL and pembrolizumab. It will also assess the antitumor efficacy and pharmacokinetics of the combination therapy compared to Lutetium (177Lu) DGUL monotherapy.

Participants will:

Monotherapy: Receive Lutetium (177Lu) DGUL 4 times (plus 2 additional doses) at 6-week intervals

Combination therapy: Receive Lutetium (177Lu) DGUL 4 times (plus 2 additional doses) at 6-week intervals along with pembrolizumab up to 18 times at 6-week intervals

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 19 years or older.
* Patients with histopathologically or cytologically confirmed adenocarcinoma of the prostate, without neuroendocrine or small cell differentiation, who have metastatic disease documented by bone lesions/soft tissue lesions and are not eligible for curative treatment.
* Patients with serum testosterone levels meeting castration levels (< 50 ng/dL) at the screening visit.
* Patients must have experienced disease progression following treatment for mCRPC with a second-generation androgen receptor signaling inhibitor therapy (e.g., abiraterone or enzalutamide).
* Docetaxel treatment is allowed for localised prostate cancer and at mHSPC stage if more than 12 months have elapsed from the last dose of docetaxel, as long as no signs of failure or disease progression occurred during or immediately after such treatment.
* Patients must be receiving hormone deprivation therapy limited to the use of LHRH agonists or LHRH antagonists throughout the study. For patients who have not undergone bilateral orchiectomy, medical castration with an LHRH agonist or antagonist must have been initiated at least 4 weeks prior to baseline and must be maintained for the entire study duration.
* Patients with prostate specific membrane antigen (PSMA)-positive disease, with a maximum standardized uptake value (SUVmax) of at least 20 at a site of disease and greater than 10 at other disease sites measuring ≥ 10mm in longest diameter.
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
* Patients with a life expectancy of at least 6 months.
* Patients with adequate hematologic, renal, and liver function, confirmed by the following criteria:

  * Absolute neutrophil count (ANC) ≥ 1,500/μL (without granulocyte colony stimulating factor (G-CSF) administration within 2 weeks prior to baseline)
  * Platelet count ≥ 100,000/μL (without transfusion within 2 weeks prior to baseline)
  * Hemoglobin ≥ 9.0 g/dL (without transfusion within 4 weeks prior to baseline)
  * Serum creatinine ≤ 1.8 mg/dL or Cockcroft-Gault creatinine clearance (CrCl) formula > 40 ml/min
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal (ULN), or ≤ 5 times the ULN for patients with confirmed liver metastasis
  * Total bilirubin ≤ 1.5 times ULN (except in patients with Gilbert syndrome)
  * Prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN
* Patients who have AEs due to previous anticancer therapies must have recovered to ≤ Grade 1 or baseline. Patients with endocrine-related AEs who are adequately treated with hormone replacement or patients who have ≤ Grade 2 neuropathy are eligible.
* Patients who voluntarily agree to participate in the clinical trial and sign the informed consent form.

Exclusion Criteria:

* Known additional malignancy that is progressing or has required active treatment within the past 3 years (Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded).
* Patients who have received chemotherapy, biological therapy, or immunotherapy for prostate cancer within 4 weeks from baseline (6 weeks in the case of nitrosoureas or mitomycin).
* Any prior treatment with taxane chemotherapy for mCRPC.
* Patients with history of allogeneic stem cell transplantation (alloSCT), or solid organ transplantation.
* Patients who have received high-dose chemotherapy requiring hematopoietic stem cell treatment, within 2 years from baseline.
* Patients who have previously received PSMA-targeted treatment (e.g., radiotherapy, immunotherapy, or antibody-drug conjugate) or those treated with radiopharmaceuticals such as radium-223 within 6 months from baseline.
* Patients who have previously received radiotherapy (RT) to the lung > 30 Gy within 6 months of the first dose.
* Prior exposure to any anti-programmed cell death protein 1(PD-1), anti-programmed death ligand 1/2 (PD-L1/L2), or anti- cytotoxic T lymphocyte antigen-4 (CTLA-4) antibody, or any other agent specifically targeting T cell co-stimulation or immune checkpoint pathways.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may enroll if they are radiologically stable (i.e., without evidence of progression) for at least 4 weeks, as confirmed by repeat imaging during the study screening. They must also be clinically stable and must not have required steroid treatment for at least 4 weeks before receiving the first dose of the study intervention.
* Patients with the following medical history or history of surgery/procedures:

  * Deep vein thrombosis (DVT) or pulmonary embolism (PE) within 1 year from baseline.
  * Cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection within 6 months from baseline.
  * Acute coronary syndrome (unstable angina or myocardial infarction) within 6 months from baseline.
  * Major cerebrovascular disease, such as stroke, within 6 months from baseline.
  * General anesthesia or major surgery requiring respiratory assistance within 4 weeks from baseline (video-assisted thoracoscopic surgery or open-and-closed (ONC) surgery allowed within 2 weeks).
  * Active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid).
  * History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Patients with the following conditions:

Class III or IV heart failure according to the New York Heart Association (NYHA) classification.

* Uncontrolled hypertension (systolic blood pressure (SBP) > 160 mm Hg or diastolic blood pressure (DBP) > 90 mm Hg).
* Clinically significant cardiovascular abnormalities as determined by the investigator (e.g., Left ventricular ejection fraction (LVEF) < 50%, clinically significant heart wall abnormalities, myocardial injury or QT interval corrected by Fridericia's formula (QTcF) > 450 msec for males or > 460 msec for females).
* Uncontrolled cardiac arrhythmia.
* Known positive human immunodeficiency virus (HIV) test or other uncontrolled active infectious diseases (e.g., Hepatitis B/C).
* Myelodysplastic syndrome (MDS).
* Clinically significant urinary obstruction or hydronephrosis that may affect renal function as determined by the investigator.

  * Patients receiving nephrotoxic drugs (e.g., aminoglycosides).
  * Patients with severe claustrophobia not controlled by anxiolytics.
  * Patients with hypersensitivity to any components of the investigational product (IP)s.
  * Patients unwilling to use appropriate contraceptive methods or abstain from intercourse during the clinical trial and for at least 4 months after discontinuation of the IPs if the patient's partner is capable of childbearing, or who do not agree to refrain from sperm donation during this period.
  * Patients who have received other IPs or undergone procedures involving investigational medical devices within 4 weeks from baseline.
  * Any other conditions deemed by the investigator as making the patient ineligible for clinical trial participation.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-emergent adverse events (TEAEs) | From enrollment to 6-month follow-up after the end of treatment
Number of patients with drug-related TEAEs | From enrollment to 6-month follow-up after the end of treatment
Adverse events (AEs) | From enrollment to 6-month follow-up after the end of treatment
Drug-related adverse reactions based on dose limited toxicity (DLT) definitions | From enrollment to 6-month follow-up after the end of treatment

SECONDARY OUTCOMES:
Radiographic progression-free survivla (rPFS) | From enrollment to 6-month follow-up after the end of treatment
1-year overall survivla (OS) | From enrollment to 6-month follow-up after the end of treatment
Objective response rate (ORR; confirmed complete response (CR) + partial response (PR)) | From enrollment to 6-month follow-up after the end of treatment
Prostate specific antigen (PSA) response rate (>50% decrease compared to baseline PSA) | From enrollment to 6-month follow-up after the end of treatment
PSA PFS | From enrollment to 6-month follow-up after the end of treatment
Best PSA response through waterfall plot | From enrollment to 6-month follow-up after the end of treatment
Disease control rate (DCR) | From enrollment to 6-month follow-up after the end of treatment
Duration of response (DOR) | From enrollment to 6-month follow-up after the end of treatment
Tumor change rate (target lesion) through waterfall plot | From enrollment to 6-month follow-up after the end of treatment
Pain severity (numeric rating scale, NRS) and opioid analgesic use | From enrollment to 6-month follow-up after the end of treatment
Quality of Life Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | From enrollment to 6-month follow-up after the end of treatment
  The EORTC QLQ-C30 measures global health status, functional scales, and symptom scales. All scores range from 0 to 100.
  For functional and global health scales, higher scores indicate better functioning.
  For symptom scales, higher scores indicate worse symptoms.
Quality of Life Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Prostate Cancer Module (EORTC QLQ-PR25) | From enrollment to 6-month follow-up after the end of treatment
  The EORTC QLQ-PR25 assesses urinary, bowel, hormonal treatment-related symptoms and sexual functioning.
  Scores range from 0 to 100. For symptom scales, higher scores indicate worse symptoms. For sexual functioning, higher scores indicate better functioning.
Quality of Life Assessed by the EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) | From enrollment to 6-month follow-up after the end of treatment
  The EQ-5D-5L generates an index value reflecting health status, typically ranging from less than 0 (worse than death) to 1 (full health).
  Higher scores indicate better overall health. A Visual Analog Scale (0-100) may also be reported, where higher scores indicate better self-rated health.
Time-Activity Curve for Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  The time-activity curve will be generated using serial imaging to quantify radioactivity kinetics of Lutetium (177Lu) DGUL in target tissues. Activity is measured in megabecquerels (MBq) over time.
Cumulative Activity of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  Cumulative activity represents the total integrated activity (MBq·h) within organs or lesions over time, derived from the time-activity curve.
Residence Time of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  Residence time is the time-integrated activity coefficient describing the average time (hours) that Lutetium (177Lu) DGUL remains in specific organs or lesions.
Effective Dose of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  The effective dose will be calculated using organ residence times and standard dosimetry models. Effective dose is reported in millisieverts (mSv).
Area Under the Plasma Concentration-Time Curve (AUC) of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  AUC represents the total systemic exposure to Lutetium (177Lu) DGUL over time. Reported in MBq·h or ng·h/mL depending on analytical method.
Peak Plasma Concentration (Cmax) of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  Cmax is the highest observed plasma concentration of Lutetium (177Lu) DGUL. Reported in MBq/mL or ng/mL.
Time to Peak Plasma Concentration (Tmax) of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  Tmax is the time at which Cmax occurs. Reported in hours.
Elimination Half-Life (T1/2) of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  T1/2 represents the time required for the plasma concentration of Lutetium (177Lu) DGUL to decrease by 50%. Reported in hours.
Volume of Distribution (Vd) of Lutetium (177Lu) DGUL | Dosimetry of Lutetium (¹⁷⁷Lu) DGUL could have a time frame of "0, 30 minutes, 1, 2, 4, 6, 24, 48, 72, and 120 hours post-dose
  Vd is the apparent volume in which Lutetium (177Lu) DGUL is distributed throughout the body. Reported in liters (L).